CLINICAL TRIAL: NCT02947256
Title: Laparoscopic Cholecystectomy With Retro-infundibular Approach Versus Standard Laparoscopic Cholecystectomy in Difficult Cases, Where Calot's Triangle is Unsafe to be Dissected
Brief Title: Laparoscopic Cholecystectomy With Retro-infundibular Approach
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, MD, Lecturer & consultant of general surgery, Department of surgery, Minia university hospital, Egypt, Minia University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fac.med.011
Record Dates: First submitted 2016-10-22; First posted 2016-10-27 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Gallstones
MeSH Terms: conditions — Gallstones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard laparoscopic cholecystectomy (Active Comparator): This included the classic dissection of Calot's triangle to achieve the CVS, with separate clipping and division of cystic duct and artery.
  Interventions: Procedure: standard laparoscopic cholecystectomy
- RI approach (Experimental): Retroinfundibular laparoscopic cholecystectomy: This included separation of the lower third of GB from its bed down to its pedicle (artery and duct) with mass ligation of both.
  Operative procedure of by RI approach:
  Interventions: Procedure: RI approach

INTERVENTIONS:
Procedure: standard laparoscopic cholecystectomy — which included the classic dissection of Calot's triangle to achieve the CVS, with separate clipping and division of cystic duct and artery
  Other Names: SLC
  Arms: standard laparoscopic cholecystectomy
Procedure: RI approach — which included separation of the lower third of GB from its bed down to its pedicle (artery and duct) with mass ligation of both.
  Arms: RI approach

SUMMARY:
Aimed to evaluate laparoscopic cholecystectomy by retro-infundibular (RI) approach compared to standard laparoscopic cholecystectomy (SLC) in difficult cases with scarred chole-cystohepatic (Calot's) triangle.

DETAILED DESCRIPTION:
This study is a prospective cohort study, conducted in Minia university hospital and Minia insurance hospital in the period from July 2013 to January 2016, where 597 patients with gallstones were admitted for laparoscopic cholecystectomy and were done by the same surgeon. Based on the preoperative scoring system to predict the degree of difficulty in laparoscopic cholecystectomy, patients that had the score > 6 and were fit for laparoscopic surgery were included in the study. Only 125 met these criteria and agreed to share in the study and gave their informed consent. 60 patients were operated by SLC (Group 1).This included the classic dissection of Calot's triangle to achieve the CVS, with separate clipping and division of cystic duct and artery. While, 65 patients were operated by laparoscopic cholecystectomy using RI approach (Group 2). This included separation of the lower third of GB from its bed down to its pedicle (artery and duct) with mass ligation of both.

Operative procedure of by RI approach:

The site of trocars was the same as for the standard cholecystectomy. After dissection of adhesion masking the GB, if present, to reach the Hartmann pouch, at this point Calot's triangle usually was scarred and frozen, the surgeon never tried to dissect it and instead the surgeon continued as follow :

1. De-shouldering of GB: by incising the serosal covering on either side of the infundibulum and lower part of the body.
2. This followed by dissection and separation of the lower third of GB body from its bed, using suction-irrigation probe or hook dissector. Dissection continued downward till the GB pedicle (duct and artery).
3. Mass ligation of cystic artery and duct, using intracorporeal note by vicryl number 1 suture.
4. Then the surgeon cut above the ligature using diathermy on scissor or ultrasound sealing device. During this step the cut end of the GB was grasped by forceps trying to prevent spillage of its content, if happened, stones were collected in a bag and extracted.
5. Then GB was dissected from its bed as usual and extracted in a bag. In cases where the GB was hugely distended, it was aspirated firstly to facilitate its grasping. Also in cases of Mirizzi syndrome the GB was opened direct on the stone to remove it, to facilitate grasping of GB then we continued as described above

ELIGIBILITY:
Inclusion Criteria:

* patient with gallstones
* score difficulty according to Gupta et al 2013 > 6
* patient fit for laparoscopic surgery

Exclusion Criteria:

* score difficulty according to Gupta et al 2013 > 6
* patient unfit for laparoscopic surgery
* refusal to share in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-07; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
conversion to open | 24 hours
  the incidence of conversion to open
biliary injury | 2 weeks
  the incidence of biliary injury

SECONDARY OUTCOMES:
operative time | 24 hours
  time from skin opening to skin closure
hospital stay | 6 weeks
  time of hospital stay
mortality | 6 weeks
  incidence of operative related mortality

CONTACTS AND LOCATIONS:
Overall Officials: Alaa M Sewefy, MD, Principal Investigator — Lecturer & consultant of general surgery, Department of surgery, Minia university hospital, Egypt.
Locations (2):
- Egypt (2):
  - Faculty of medicine, Minya
  - Minia University Hospital, Minya

IPD SHARING:
Plan to Share IPD: No